CLINICAL TRIAL: NCT03437031
Title: Virtual Reality in Labor and Delivery for Reduction in Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with recruitment
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Gregory, Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050082
Record Dates: First submitted 2018-01-16; First posted 2018-02-19 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Labor Pain; Virtual Reality; Alternative Medicine
Keywords: Labor Pain; Virtual Reality; Alternative Medicine
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Latent-Control (No Intervention): Patients in the latent phase of labor who will receive no intervention.
- Latent-Virtual Reality (VR) (Experimental): Patients in the latent phase of labor who will receive the Virtual Reality (VR) intervention.
  Interventions: Device: Virtual Reality device

INTERVENTIONS:
Device: Virtual Reality device — For those patients randomized to VR, the study staff member will explain the use of the Samsung VR goggle set, and thereafter will allow the patient to use the device freely for up to 30 minutes. Intervals of 2-5 minutes is suggested for first-time use, and patients will be to allowed to discontinue it at any time as long as they are not experiencing any discomfort or side effects (dizziness, motion sickness, etc.). The study staff member will be present at all times, and will work with hospital staff as necessary to ensure the patient is receiving appropriate clinical care throughout the duration of the intervention.
  Arms: Latent-Virtual Reality (VR)

SUMMARY:
The purpose of this study is to identify whether use of virtual reality devices can improve the pain management of women in labor and delivery. The investigators will perform a randomized controlled trial of patients in labor at Cedars-Sinai Medical Center.

DETAILED DESCRIPTION:
The purpose of this study is to identify whether use of virtual reality devices can improve the pain management of women in labor and delivery. The investigators hypothesize that use of virtual reality devices will result in a reduction in pain medication use, in epidural use, and prolong the duration of time prior to the patient receiving an epidural.

The study will be conducted as two parallel randomized controlled trials: one for latent labor patients and one for patients in active labor (defined by whether they are < 6 cm or > 6 cm). Within each phase of labor, there will be 20 in the Virtual Reality arm and 20 in the Control arm for a total of 80 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. >18 years old
3. Pregnant with term gestation
4. Nullipara
5. Pain due to contractions rated from 4-7
6. Contractions at least every 5 minutes x 30 minutes preceding
7. Pain scores obtained at least every 60 minutes

Exclusion Criteria:

1. Parous
2. Use of intravenous medications for pain relief prior to the intervention
3. Use of an epidural
4. Preterm gestation
5. Pain not due to contractions
6. Pain score of 3 or below or 8 or above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in March 2018 and completed in February 2019. Patients were recruited in the labor and delivery inpatient setting.
Pre-assignment Details: No events occurred between recruitment, enrollment, and randomization/assignment to a study arm.
Groups:
- Latent-VR: Patients in the latent phase of labor who will receive the VR intervention.
  Virtual Reality device: For those patients randomized to VR, the study staff member will explain the use of the Samsung VR goggle set, and thereafter will allow the patient to use the device freely for up to 30 minutes. Intervals of 2-5 minutes is suggested for first-time use, and patients will be to allowed to discontinue it at any time as long as they are not experiencing any discomfort or side effects (dizziness, motion sickness, etc.). The study staff member will be present at all times, and will work with hospital staff as necessary to ensure the patient is receiving appropriate clinical care throughout the duration of the intervention.
Period: Overall Study
Arm/Group | Latent-Control | Latent-VR
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Active-Control and Active-VR participants were not recruited
Groups:
- Total: Total of all reporting groups
Arm/Group | Latent-Control | Latent-VR | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Full Range); unit: years] | 32.47 [27 to 42] | 31.57 [20 to 39] | 32 [20 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 18 | 15 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 14 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Gravidity [Mean (Full Range); unit: pregnancies] | 1.16 [1 to 3] | 1.29 [1 to 3] | 1.23 [1 to 3]
Parity [Mean (Full Range); unit: pregnancies] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Insurance [Count of Participants; unit: Participants]
  HMO / Managed Care | 0 | 4 | 4
  Medicaid | 1 | 2 | 3
  Private | 18 | 14 | 32
  Self-pay / None | 0 | 1 | 1
BMI [Mean (Full Range); unit: kg/m^2] | 27.29 [22.5 to 38.4] | 30.11 [24.1 to 38.6] | 28.77 [22.5 to 38.6]

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Pain
Description: Difference in pain scores pre-post intervention compared to control. The investigators will use the Visual Analog Scale (VAS) for Pain. The minimum pain is 1; the maximum is 10. Higher values represent more pain.
Time Frame: 4 hours prior to intervention, immediately pre-intervention, immediately post-intervention, 2, 4, 24 hours post-intervention
Population: Average Pain Score in 2 hours AFTER Intervention data available only for 9/19 Latent-Control participants and 14/21 Latent-VR participants Average Pain Score in 4 hours AFTER Intervention data available only for 7/19 Latent-Control participants and 12/21 Latent-VR participants Average Pain Score in 24 hours AFTER Intervention data available only for 0/19 Latent-Control participants and 2/21 Latent-VR participants
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Latent-Control | Latent-VR
Number analyzed (Participants) | 19 | 21
score on a scale
  Average Pain Score in 4 hours PRIOR to Intervention | 3.39 [0 to 7] | 4.52 [1.3 to 7]
  Pre-Intervention Pain score | 5.05 [4 to 7] | 6 [4 to 7]
  Post-Intervention Pain score | 5.63 [4 to 10] | 5.48 [0 to 8]
  Average Pain Score in 2 hours AFTER Intervention: number analyzed (Participants) | 9 | 14
  Average Pain Score in 2 hours AFTER Intervention | 5.44 [4 to 7.5] | 5 [0 to 8]
  Average Pain Score in 4 hours AFTER Intervention: number analyzed (Participants) | 7 | 12
  Average Pain Score in 4 hours AFTER Intervention | 6.2 [4.3 to 8.7] | 5.48 [1 to 8.5]
  Average Pain Score in 24 hours AFTER Intervention: number analyzed (Participants) | 0 | 2
  Average Pain Score in 24 hours AFTER Intervention |  | 3.36 [2.75 to 4]

2. Secondary Outcome: Number of Participants With a Need for Intravenous Pain Medication
Description: IV pain medication during the intervention (yes/no)
Time Frame: The total duration of the intervention (30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Latent-Control | Latent-VR
Number analyzed (Participants) | 19 | 21
Participants | 0 | 0

3. Secondary Outcome: Need for Epidural During the Intervention
Description: Number of participants with need for an epidural during the intervention
Time Frame: The total duration of the intervention (30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Latent-Control | Latent-VR
Number analyzed (Participants) | 19 | 21
Participants | 0 | 0

4. Secondary Outcome: Childbirth Self-Efficacy Inventory
Description: The Childbirth Self-Efficacy Inventory (CSEI) is a measure of how well a patient anticipates being able to perform certain tasks in labor such as relaxing their body, keeping calm, or not thinking about the pain. The investigators will ask to what extend they feel virtual reality would be able to influence their ability to do these things. A fifteen-question scale reflecting degree of control where 1 is least control and 5 is most control per item. Minimum score 15 reflecting least total control; maximum score 75 reflecting maximal control.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Latent-Control | Latent-VR
Number analyzed (Participants) | 19 | 21
score on a scale | 54.8 (11.2) | 52.6 (11.8)

5. Secondary Outcome: Number of Participants With a Need for Epidural During the Labor
Description: Epidural use during labor (yes/no)
Time Frame: The total duration of the patient's labor (average 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Latent-Control | Latent-VR
Number analyzed (Participants) | 19 | 21
Participants | 17 | 18

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: 0 participants in Active-Control group and 0 participants Active-VR group. Participants were not recruited into these two groups.
Groups:
- Active-Control: Patients in the active phase of labor who will receive no intervention.
- Active-VR: Patients in the active phase of labor who will receive the VR intervention.
  Virtual Reality device: For those patients randomized to VR, the study staff member will explain the use of the Samsung VR goggle set, and thereafter will allow the patient to use the device freely for up to 30 minutes. Intervals of 2-5 minutes is suggested for first-time use, and patients will be to allowed to discontinue it at any time as long as they are not experiencing any discomfort or side effects (dizziness, motion sickness, etc.). The study staff member will be present at all times, and will work with hospital staff as necessary to ensure the patient is receiving appropriate clinical care throughout the duration of the intervention.
Arm/Group | Latent-Control | Latent-VR | Active-Control | Active-VR
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03437031/Prot_SAP_001.pdf